CLINICAL TRIAL: NCT01459835
Title: Media Impact on Preschool Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Dimitri Christakis, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01HD056506-02 (NIH)
Record Dates: First submitted 2011-10-21; First posted 2011-10-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Aggression; Prosocial Behavior
Keywords: TV; Violence; DVDs; Behavior; Preschool children
MeSH Terms: conditions — Aggression; Altruism; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- media diet (Experimental): advice tips and tools to reduce exposure to violent programming
  Interventions: Behavioral: media diet
- Nutrition intervention (Active Comparator): diet advice
  Interventions: Behavioral: nutritional intervention

INTERVENTIONS:
Behavioral: media diet — advice and tips and tools for healthy non violent TV viewing
  Arms: media diet
Behavioral: nutritional intervention — advice on healthy eating
  Arms: Nutrition intervention

SUMMARY:
This study tests the hypothesis that modifying the media diet of preschool children so that they watch more prosocial programming and less violent programming will result in decreased aggression and increased prosocial behavior.

ELIGIBILITY:
Inclusion Criteria:

* 2.5-4 years of age
* watches TV regularly
* English speaking

Exclusion Criteria:

* no TV
* non English

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Social Competence and Behavioral Evaluation (SCBE) scores overall | 6 months after enrollment
  Overall Social Competence and Behavioral Evaluation (SCBE) scores will be assessed
Social Competence and Behavioral Evaluation (SCBE) aggression subscale | 6 months after enrollment
  Aggression, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed at 6,
Social Competence and Behavioral Evaluation (SCBE) prosocial subscale | 6 months after enrollment
  Prosocial, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed
Social Competence and Behavioral Evaluation (SCBE) scores overall | 12 months after enrollment
  Overall Social Competence and Behavioral Evaluation (SCBE) scores will be assessed
Social Competence and Behavioral Evaluation (SCBE) scores overall | 18 months after enrollment
  Overall Social Competence and Behavioral Evaluation (SCBE) scores will be assessed
Social Competence and Behavioral Evaluation (SCBE) aggression subscale | 12 months after enrollment
  Aggression, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed
Social Competence and Behavioral Evaluation (SCBE) aggression subscale | 18 months after enrollment
  Aggression, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed
Social Competence and Behavioral Evaluation (SCBE) prosocial subscale | 12 months after enrollment
  Prosocial, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed
Social Competence and Behavioral Evaluation (SCBE) prosocial subscale | 18 months after enrollment
  Prosocial, from the Social Competence and Behavioral Evaluation (SCBE) subscale scores, will be assessed

SECONDARY OUTCOMES:
sleep problems | 6 months
  The investigator will use elements of the sleep problem questionnaire to assess sleep problems
sleep problems | 12 months
  The investigator will use elements of the sleep problem questionnaire to assess sleep problems
sleep problems | 18 months
  The investigator will use elements of the sleep problem questionnaire to assess sleep problems

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Christakis, MD, Principal Investigator — U of WA
Locations (1):
- Seattle CHildrens Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Christakis DA, Garrison MM, Herrenkohl T, Haggerty K, Rivara FP, Zhou C, Liekweg K. Modifying media content for preschool children: a randomized controlled trial. Pediatrics. 2013 Mar;131(3):431-8. doi: 10.1542/peds.2012-1493. Epub 2013 Feb 18. PMID 23420911
- [Derived] Garrison MM, Christakis DA. The impact of a healthy media use intervention on sleep in preschool children. Pediatrics. 2012 Sep;130(3):492-9. doi: 10.1542/peds.2011-3153. Epub 2012 Aug 6. PMID 22869826